CLINICAL TRIAL: NCT07331428
Title: Efficacy and Safety of MRG003 With PD-1 Induction Followed by Capecitabine and PD-1 Maintenance as First-line Treatment in Locally Recurrent Nasopharyngeal Carcinoma
Brief Title: MRG003 Induction and Capecitabine Maintenance With PD-1 in Locally Recurrent NPC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qiaojuan Guo, PhD, Fujian Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-12-19
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Nasopharyngeal Carcinoma; Local Recurrence
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — tislelizumab; Capecitabine

STUDY DESIGN:
Intervention Model Description: The treatment regimen includes an induction phase with MRG003 at 2.0 mg/kg (D1) combined with Tislelizumab 200 mg (D1), administered weekly for 6 cycles. This is followed by maintenance therapy consisting of Capecitabine (650 mg/m², twice daily on days 1-21) in combination with Tislelizumab, continued for up to 1 year or until disease progression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRG003 (Experimental): The treatment regimen comprises an induction phase with MRG003 at 2.0 mg/kg (administered on Day 1) in combination with Tislelizumab 200 mg (also on Day 1), delivered every three weeks for a total of six cycles. Upon achieving an objective response (ORR), patients will proceed to maintenance therapy, which consists of Capecitabine (650 mg/m², administered twice daily on Days 1-21) in conjunction with Tislelizumab. This maintenance phase will continue for up to one year or until disease progression is observed.
  Interventions: Drug: MRG003; Drug: Tislelizumab; Drug: Capecitabine

INTERVENTIONS:
Drug: MRG003 — MRG003 at 2.0 mg/kg (D1) will be administered every three weeks for 6 cycles
Drug: Tislelizumab — Tislelizumab 200 mg (D1) will be administered every three weeks for 6 cycles. Upon achieving an objective response, maintenance therapy will continue for up to one year or until disease progression is observed.
Drug: Capecitabine — After achieving an objective response (ORR) with the combination of MRG003 and Tislelizumab, maintenance therapy will consist of Capecitabine (650 mg/m², administered twice daily on Days 1-21) in conjunction with Tislelizumab. This maintenance phase will continue for up to one year or until disease progression is observed.

SUMMARY:
This study enrolls patients who have experienced local recurrence of nasopharyngeal carcinoma (NPC) with or without regional recurrence. The treatment regimen includes an induction phase with MRG003 at 2.0 mg/kg (D1) combined with Tislelizumab 200 mg (D1), administered weekly for 6 cycles. This is followed by maintenance therapy consisting of Capecitabine (650 mg/m², twice daily on days 1-21) in combination with Tislelizumab, continued for up to 1 year or until disease progression.

ELIGIBILITY:
Inclusion Criteria:

**Inclusion Criteria:**

1. Patients with locally recurrent nasopharyngeal carcinoma (NPC) more than 1 year after initial radical treatment for non-metastatic NPC, with or without regional recurrence, but without distant metastasis.
2. Age 18-70 years.
3. Pathologically confirmed local recurrence of NPC, staged as rT1-rT4 according to the 9th edition of the AJCC/UICC classification.
4. ECOG performance status score of 0-1.
5. No prior radiotherapy, chemotherapy, immunotherapy, or biological therapy for recurrent NPC.
6. No contraindications to immunotherapy or chemotherapy.
7. Adequate organ function.

Exclusion Criteria:

**Exclusion Criteria:**

1. Previous treatment with other PD-1 antibodies or immunotherapy targeting PD-1/PD-L1 resulting in Grade III or higher immune-related adverse reactions.
2. Residual toxic effects from prior anti-tumor treatments (including immunotherapy, targeted therapy, chemotherapy, or radiotherapy) (excluding alopecia, fatigue, and Grade 2 hypothyroidism) or clinically significant laboratory abnormalities higher than Grade 1 (CTCAE v5.0).
3. Congenital or acquired immunodeficiency (e.g., HIV infection), active hepatitis B (HBV-DNA ≥10 copies/ml), or hepatitis C (positive hepatitis C antibody and HCV-RNA above the detection limit of the assay).
4. Known allergy to MRG003, capecitabine, or any component of anti-PD-1 antibodies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Day 21 after the completion of six cycles of MRG003 treatment
  The Objective Response Rate (ORR) is defined as the proportion of patients achieving Complete Response (CR) or Partial Response (PR) by Day 21 after the completion of six cycles of MRG003 treatment, starting from the date of enrollment.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 1-year; 3-year
  PFS is defined as the time from enrollment to the date of tumor progression or death from any cause, or to the date of the last follow-up if no progression has occurred.
Overall Survival (OS) | 1-year; 3-year
  OS is defined as the time from enrollment to the date of death from any cause, or to the date of the last follow-up if no death has occurred.
Duration of Response (DOR) | 1-year; 3-year
  DOR is defined as the time from the first assessment of Complete Response (CR) or Partial Response (PR) to the first assessment of Progressive Disease (PD) or death from any cause
Disease Control Rate (DCR) | Day 21 after the completion of six cycles of MRG003 treatment
  DCR is defined as the proportion of subjects who achieve Complete Response (CR), Partial Response (PR), or Stable Disease (SD) after treatment.

IPD SHARING:
Plan to Share IPD: No